CLINICAL TRIAL: NCT01487616
Title: Prevalence of Congenital Uterine Malformations in Women With a History of Preterm Delivery or Miscarriage
Brief Title: Prevalence of Congenital Uterine Malformations
Acronym: PUMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 11072
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Congenital Uterine Anomalies
Keywords: Mullerian anomalies; Congenital uterine malformations or anomalies; Arcuate; Septate; Subseptate; Bicornuate; Unicornuate; Didelphys; T-shaped
MeSH Terms: conditions — Congenital Abnormalities; Uterine Didelphys

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Women with previous preterm birth: Women with history of preterm birth (birth of a baby of less than 37 weeks gestational age, where labour was spontaneous) regardless of past pregnancy history.
- Women with previous miscarriage: Women with history of miscarriage (spontaneous pregnancy loss before 24 weeks of gestation), regardless of past pregnancy history.
- Women with previous term births: Women with previous term births (37 or more weeks of gestation)

SUMMARY:
Aims: We plan to investigate how common uterine malformations are in high-risk women (with history of miscarriage or preterm delivery), by analysing different characteristics in these groups. This study will also investigate other ultrasound characteristics detected on these women. This study will point towards the possible mechanism of how uterine malformations may affect pregnancy outcomes.

DETAILED DESCRIPTION:
Background: Congenital abnormally shaped wombs (uterine malformations) have long been thought to be more common in women with poor pregnancy outcomes, e.g. miscarriage (Rackow and Arici 2007) and preterm delivery (Tomazevic, Ban-Frangez et al. 2007). However, the true prevalence is difficult to assess as there are no universally agreed classification systems and some of the best investigations are invasive. In addition, previous prevalence studies have not examined the details of subfertility or pregnancy loss, such as duration of subfertility, the gestation of pregnancy loss, or miscarriage pattern.

Aims: We plan to investigate how common uterine malformations are in high-risk women (with history of miscarriage or preterm delivery), by analysing different characteristics in these groups. This study will also investigate other ultrasound characteristics detected on these women. This study will point towards the possible mechanism of how uterine malformations may affect pregnancy outcomes.

Methods: We plan to recruit women who have had miscarriage or preterm delivery into our study. A sample of women who had normal term deliveries will be recruited as comparison. All women will undergo one 3-dimensional ultrasound scan each.

Outcomes: The proportions of women with congenital uterine malformations will be determined. Any ultrasound-detected markers found especially in women with poor pregnancy outcomes may point towards how uterine malformations affect pregnancies.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a previous miscarriage

   * Age: 18 years old or more
   * Definition of miscarriage: the spontaneous pregnancy loss up until 24 weeks of gestation, where the pregnancy was confirmed histologically or with previous presence of a gestational sac with or without fetal pole and fetal heart activity on ultrasound scanning.
   * At least 8 weeks after the end of last pregnancy
2. Women with preterm birth

   * Age: 18 years old or more
   * Definition of preterm birth: birth at less than 37 weeks of gestation.
   * At least 8 weeks after the end of last pregnancy
3. Control group (women with term birth)

   * Age: 18 years old or more
   * Definition of term birth: birth at 37 or more weeks of gestation
   * At least 8 weeks after the end of last pregnancy

Exclusion Criteria:

* Pregnant at the date of the 3D TVUS
* Recent uterine or endometrial surgery
* Women unable to tolerate 3D TVUS
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care: Patients from Nottingham University Hospitals NHS Trust
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Presence of uterine malformations | At least 8 weeks after the end of last pregnancy
  Presence of uterine malformations in study group compared to control group

SECONDARY OUTCOMES:
Ultrasound markers on pelvic 3D ultrasound | At least 8 weeks after the end of last pregnancy
  Ultrasound markers on pelvic 3D ultrasound in study versus control group

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Raine-Fenning, MBChB PhD, Principal Investigator — The University of Nottingham
Locations (1):
- Academic Imaging Suite, The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan YY, Jayaprakasan K, Zamora J, Thornton JG, Raine-Fenning N, Coomarasamy A. The prevalence of congenital uterine anomalies in unselected and high-risk populations: a systematic review. Hum Reprod Update. 2011 Nov-Dec;17(6):761-71. doi: 10.1093/humupd/dmr028. Epub 2011 Jun 24. PMID 21705770
- [Background] Chan YY, Jayaprakasan K, Tan A, Thornton JG, Coomarasamy A, Raine-Fenning NJ. Reproductive outcomes in women with congenital uterine anomalies: a systematic review. Ultrasound Obstet Gynecol. 2011 Oct;38(4):371-82. doi: 10.1002/uog.10056. PMID 21830244